CLINICAL TRIAL: NCT06239181
Title: The Effect of Breathing Exercises Applied to Patients Undergoing Coronary Angiography for the First Time on Anxiety
Brief Title: Effect of Breathing Exercises Before Coronary Angiography
Acronym: EBECA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Rahşan Yılmaz, Nurse, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/01-06
Record Dates: First submitted 2024-01-17; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Anxiety; Breathing Exercises
Keywords: Coronary angiography; Breathing exercises; Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: The study included 2 groups, experimental and control. The patients in the experimental group were administered the beck anxiety scale before coronary angiography. the patients in the experimental group were given breathing exercises by the researcher for 15-20 minutes. the beck anxiety scale was reapplied after the procedure. the patients in the control group were not administered any application and the beck anxiety scale was reapplied after the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EBECA (Experimental): The patients in the intervention group scheduled for angiography were administered the Beck Anxiety Scale, and then they underwent conscious, deep breathing exercises along with synchronized breathing training. The face-to-face teaching and application of the breathing exercises took an average of 15-20 minutes.
  Interventions: Behavioral: Breathing Exercises
- control group (Active Comparator): For the patients in the control group who were scheduled for angiography, the Beck Anxiety Scale was administered face-to-face before the procedure, and they were then sent for the procedure after receiving routine treatment without any additional intervention.
  Interventions: Other: no intervention/routine procedure

INTERVENTIONS:
Behavioral: Breathing Exercises — The patients in the intervention group scheduled for angiography were administered the Beck Anxiety Scale, and then they underwent conscious, deep breathing exercises along with synchronized breathing training. The face-to-face teaching and application of the breathing exercises took an average of 15-20 minutes. Additionally, routine treatment was applied. For both the intervention and control groups, the Beck Anxiety Scale was administered again after the completion of the coronary angiography procedure, once stabilization was achieved.
  Arms: EBECA
Other: no intervention/routine procedure — Beck Anxiety Scale was administered to the control group before coronary angiography. No intervention was performed in between. The routine procedure of the hospital continued. Beck Anxiety Scale was administered again after leaving the procedure.
  Arms: control group

SUMMARY:
This research was designed as a pre-test-post-test controlled group randomized controlled interventional study to determine the effect of breathing exercises applied to patients undergoing coronary angiography for the first time on anxiety. Patients were provided with an informed consent form, a personal information form and the Beck Anxiety Scale. The Beck Anxiety Scale was administered to the control group before and after the procedure. In the experimental group, the Beck Anxiety Scale was administered before the procedure, and after providing breathing exercise education and application, the Beck Anxiety Scale was completed after the procedure.

DETAILED DESCRIPTION:
This research was designed as a pre-test-post-test controlled group randomized controlled interventional study to determine the effect of breathing exercises applied to patients undergoing coronary angiography for the first time on anxiety.

The study population consisted of SBÜ Kartal Koşuyolu Training and Research Hospital.When statistical power analysis was performed according to the G-Power program in the sample group, a minimum of 34 experimental and a minimum of 34 control groups were used, considering data loss, 76 volunteer patients who met the inclusion criteria were studied. Patients were provided with an informed consent form, a personal information form and the Beck Anxiety Scale. The Beck Anxiety Scale was administered to the control group before and after the procedure. In the experimental group, the Beck Anxiety Scale was administered before the procedure, and after providing breathing exercise education and application, the Beck Anxiety Scale was completed after the procedure. The 'Dependent Group T-Test' technique was used for the analysis of data obtained from the scales used in the study, comparing pre-test and post-test scores of the intervention and control groups. Also, the 'Independent Group T-Test' was used for separate comparisons of pre-test and post-test scores of the experimental and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Were between 18-80 years old,
* Had never undergone coronary angiography before,
* Correctly and completely filled out the Beck Anxiety Scale,
* Voluntarily agreed to participate in the study.

Exclusion Criteria:

* Having a psychiatric illness
* Communication problems

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Beck Anxiety Inventory | 1 year
  Patients who completed the Beck Anxiety Inventory were evaluated based on the scores they provided. The options were scored as follows: 'Not at all' option received 0 points, 'Mild' received 1 point, 'Moderate' received 2 points, and 'Severe' received 3 points. Scores were totaled at the end of the test. The evaluation was explained as follows:
  8-15 points = Mild anxiety level 16-25 points = Moderate anxiety level 26-63 points = Severe anxiety level

CONTACTS AND LOCATIONS:
Locations (1):
- Maltepe University, Maltepe, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided